CLINICAL TRIAL: NCT03695601
Title: Surveillance HeartCare® Outcomes Registry
Acronym: SHORE
Status: Active, not recruiting | Type: Observational
Sponsor: CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: SN-C-00011
Record Dates: First submitted 2018-09-28; First posted 2018-10-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Heart Transplant Rejection
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For AlloMap, RNA isolated from peripheral blood mononuclear cells (PBMC) For AlloSure-Heart, plasma from venous blood will be collected and cell-free DNA will be extracted from the plasma for analysis of donor-derived cell-free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HeartCare: Diagnostic Test: Heart Care 2300 patients managed with HeartCare (AlloMap® and AlloSure-Heart® )
  Interventions: Other: Standard of Care
- Control: A historical control group will be matched to the estimated 1150 HeartCare group patients who complete at least two years of HeartCare surveillance use and inclusive of year 3 post-transplant clinical follow-up for outcome. The criteria for the matched controls will be based on allograft donor type, age, gender, ethnicity/race, and other clinical factors. Propensity scores will be used to perform the matching.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Other Standard measures for monitoring rejection: Endomyocardial Biopsy, Echocardiogram, Angiography, Intravascular Ultrasound, Donor-specific HLA Antibody

SUMMARY:
This is an observational registry to assess the clinical utility of surveillance using HeartCare testing services, in association with clinical care of heart transplant recipients.

DETAILED DESCRIPTION:
HeartCare is a service which includes AlloMap® and AlloSure-Heart® to provide information to help clinicians to more comprehensively monitor heart transplant recipients for allograft rejection. An approach to surveillance using HeartCare provides information from two complementary measures; AlloMap is a gene-expression profile based measure of host immune activity and risk of acute rejection. AlloSure-Heart monitors graft injury. AlloMap is the first FDA cleared test and is the only non-invasive, blood test method recommended in the International Society for Heart and Lung Transplantation (ISHLT) guidelines for surveillance of heart transplant recipients for rejection. AlloSure-Heart measures donor-derived cell-free DNA (dd-cfDNA) to help discriminate acute cellular rejection and antibody-mediated rejection from no rejection. Patients who receive HeartCare, as part of their post-transplant management, will give informed consent for information on their outcomes and other relevant clinical information, found in their medical records, to be entered into a SHORE database for purposes of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 15 years of age or older at the time of blood draw.
2. Received a heart transplant (primary or repeat)
3. Patients who have HeartCare initiated within 3 months post-transplant

Exclusion Criteria:

1. Patients who are pregnant at the time of blood draw.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible heart transplant recipients who meet the inclusion/exclusion criteria will be a part of this observational study.
  The control cohort will include the historical patients cared for without the use of HeartCare at the participating centers.
Sampling Method: Probability Sample
Enrollment: 2743 (Estimated)
Dates: Start 2018-12-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who develop de-novo DSA as a surrogate to clinical outcomes at 1, 3 and 5 years post-transplant. | Dec-2026
  The primary endpoint of the study is the proportion of patients who develop de-novo DSA as a surrogate to clinical outcomes at 1, 3 and 5 years post-transplant. The overall incidence of de-novo DSA is between 10-20% in the first year and 10-15% each year subsequently.

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Khush, MD, Principal Investigator — Stanford University
Locations (67):
- United States (67):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Baptist Health Arkansas, Little Rock, Arkansas
  - University of California San Diego, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - University of California San Fransisco Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - Yale New Haven, New Haven, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Memorial Healthcare System, Hollywood, Florida
  - Mayo Clinic- Florida, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Advent Health, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Ascension St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Barnes Jewish Hospital, Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Northwell Health/ North Shore University Hospital, Manhassett, New York
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - Saint Thomas Health, Nashville, Tennessee
  - Ascension Seton, Austin, Texas
  - Medical City Dallas, Dallas, Texas
  - Baylor Research Institute, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - UTHealth/ Memorial Hermann Hospital, Houston, Texas
  - Methodist Healthcare Systems of San Antonio, San Antonio, Texas
  - Intermountain Heart Institute, Murray, Utah
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Research Institute, Milwaukee, Wisconsin

REFERENCES:
- [Background] Agbor-Enoh S, Tunc I, De Vlaminck I, Fideli U, Davis A, Cuttin K, Bhatti K, Marishta A, Solomon MA, Jackson A, Graninger G, Harper B, Luikart H, Wylie J, Wang X, Berry G, Marboe C, Khush K, Zhu J, Valantine H. Applying rigor and reproducibility standards to assay donor-derived cell-free DNA as a non-invasive method for detection of acute rejection and graft injury after heart transplantation. J Heart Lung Transplant. 2017 Sep;36(9):1004-1012. doi: 10.1016/j.healun.2017.05.026. Epub 2017 May 20. PMID 28624139
- [Background] Crespo-Leiro MG, Stypmann J, Schulz U, Zuckermann A, Mohacsi P, Bara C, Ross H, Parameshwar J, Zakliczynski M, Fiocchi R, Hoefer D, Colvin M, Deng MC, Leprince P, Elashoff B, Yee JP, Vanhaecke J. Clinical usefulness of gene-expression profile to rule out acute rejection after heart transplantation: CARGO II. Eur Heart J. 2016 Sep 1;37(33):2591-601. doi: 10.1093/eurheartj/ehv682. Epub 2016 Jan 7. PMID 26746629
- [Background] De Vlaminck I, Valantine HA, Snyder TM, Strehl C, Cohen G, Luikart H, Neff NF, Okamoto J, Bernstein D, Weisshaar D, Quake SR, Khush KK. Circulating cell-free DNA enables noninvasive diagnosis of heart transplant rejection. Sci Transl Med. 2014 Jun 18;6(241):241ra77. doi: 10.1126/scitranslmed.3007803. PMID 24944192
- [Background] Deng MC, Eisen HJ, Mehra MR, Billingham M, Marboe CC, Berry G, Kobashigawa J, Johnson FL, Starling RC, Murali S, Pauly DF, Baron H, Wohlgemuth JG, Woodward RN, Klingler TM, Walther D, Lal PG, Rosenberg S, Hunt S; CARGO Investigators. Noninvasive discrimination of rejection in cardiac allograft recipients using gene expression profiling. Am J Transplant. 2006 Jan;6(1):150-60. doi: 10.1111/j.1600-6143.2005.01175.x. PMID 16433769
- [Background] Grskovic M, Hiller DJ, Eubank LA, Sninsky JJ, Christopherson C, Collins JP, Thompson K, Song M, Wang YS, Ross D, Nelles MJ, Yee JP, Wilber JC, Crespo-Leiro MG, Scott SL, Woodward RN. Validation of a Clinical-Grade Assay to Measure Donor-Derived Cell-Free DNA in Solid Organ Transplant Recipients. J Mol Diagn. 2016 Nov;18(6):890-902. doi: 10.1016/j.jmoldx.2016.07.003. Epub 2016 Oct 7. PMID 27727019
- [Background] Kobashigawa J, Patel J, Azarbal B, Kittleson M, Chang D, Czer L, Daun T, Luu M, Trento A, Cheng R, Esmailian F. Randomized pilot trial of gene expression profiling versus heart biopsy in the first year after heart transplant: early invasive monitoring attenuation through gene expression trial. Circ Heart Fail. 2015 May;8(3):557-64. doi: 10.1161/CIRCHEARTFAILURE.114.001658. Epub 2015 Feb 19. PMID 25697852
- [Background] Pham MX, Teuteberg JJ, Kfoury AG, Starling RC, Deng MC, Cappola TP, Kao A, Anderson AS, Cotts WG, Ewald GA, Baran DA, Bogaev RC, Elashoff B, Baron H, Yee J, Valantine HA; IMAGE Study Group. Gene-expression profiling for rejection surveillance after cardiac transplantation. N Engl J Med. 2010 May 20;362(20):1890-900. doi: 10.1056/NEJMoa0912965. Epub 2010 Apr 22. PMID 20413602
- [Derived] Kim PJ, Alam AH, Teuteberg JJ, Khush KK, Pinney SP, Cheng RK, Yehya A, Kobulnik J, Pinney KM, Oreschak KA, Ensor CR, Fan S, Urey MA, Shah P, Hall SA. Donor-Derived Cell-Free DNA in Antibody-Mediated Rejection: An Analysis of the Surveillance HeartCare Outcomes Registry. JACC Heart Fail. 2026 Jan;14(1):102716. doi: 10.1016/j.jchf.2025.102716. Epub 2025 Oct 22. PMID 41123513